CLINICAL TRIAL: NCT00662805
Title: A 2-year Observational Study to Evaluate Safety of Seretide 50/500μg Twice Daily Administered by DISKUS, in Patients With COPD
Brief Title: Pharmacovigilance Study to Evaluate Safety of SERETIDE in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 104246; Seretide-pv/GR (Other: GlaxoSmithKline)
Record Dates: First submitted 2008-04-14; First posted 2008-04-21 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: pharmacovigilance; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants will undergo physical examination and blood pressure measurement. A complete medical history will be taken, as well as blood and urine samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Salmeterol/Fluticasone propionate (50/500 μg): Open label, 6 visits, single arm study
  Interventions: Drug: Salmeterol/Fluticasone propionate

INTERVENTIONS:
Drug: Salmeterol/Fluticasone propionate — Open label, of Salmeterol/Fluticasone propionate (50/500 μg) twice daily via dry powder inhaler (DPI)

SUMMARY:
Primary objective: Evaluation of the safety of Seretide discus administration in subjects with COPD. Treatment duration: 2 years. Study has 3 phases: Screening phase (visit 1), treatment phase (visits 2-5. In the case of AE, there will be another visit (visit 6) as a follow up visit - follow up phase.

ELIGIBILITY:
Inclusion Criteria:

* Subject should fulfill criteria for the subscription of SERETIDE as these are mentioned in SPC.

Exclusion Criteria:

* Hypersensitivity to Salmeterol + Fluticasone or any of its excipients
* Pregnancy, lactation or scheduled pregnancy during the observational period of the study
* Serious illness/disease, not adequately controlled, or with a potential to interfere with the patients' participation in the present study, according to the investigator/physician's judgment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Planned: 1000 / Recruited: 771 / Analyzed: 771 A target enrolment of approximately 1000 subjects is planned, at outpatient sites. Any subject with COPD who has an indication to receive Salmeterol + Fluticasone 50/500mcg twice daily at the discretion of the investigator and has met all the inclusion criteria, may take part in the study.
  Inclusion criteria
  * Outpatient diagnosed with COPD (Criteria of the British Thoracic Society or NHLBI/WHO Global initiative for Chronic Obstructive Lung Disease)
  * FEV1 < 50% of the one predicted at treatment start and/or
  * History of repetitive COPD exacerbations and/or
  * Patient remains symptomatic despite regular bronchodilator therapy
Sampling Method: Non-Probability Sample
Enrollment: 762 (Actual)
Dates: Start 2004-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The change in markers of increased cardiovascular risk (e.g proinflammatory and prothrombotic markers, microalbuminuria) | 104 weeks
  Evaluate adverse events, vital sign reporting, and concomitant medications

SECONDARY OUTCOMES:
Trough FEV1, FVC and FEV1/ FVC ratio | every 26 weeks
Health status as determined using the St George's Respiratory Questionnaire (SGRQ) | every 26 weeks
Laboratory assessment including levels of appropriate cardiovascular markers (e.g. CRP, Fibrinogen, PAI-1) and established risk factors, as well as detection of microalbuminuria | every 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline